CLINICAL TRIAL: NCT00924547
Title: Oral Docosahexanoic Acid Supplementation in Cystic Fibrosis: Effects on Exhaled Pro-inflammatory Isoprostanes and Analysis of Its Esterification Sites in Plasma
Brief Title: Oral Docosahexanoic Acid Supplementation in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael O'Connor, Pediatric Pulmonary Fellow, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 081363
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Docosahexanoic Acid; DHA; isoprostanes; fatty acid
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docosahexanoic Acid Supplement (Experimental): In this arm, participants took two different doses of a DHA supplement. Each dose of the DHA supplement was taken for 4 weeks.
  Interventions: Dietary Supplement: Docosahexanoic Acid Supplement
- Placebo (Placebo Comparator): In this arm, participants took a placebo pill that did not contain any DHA.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexanoic Acid Supplement — The active treatment will consist of Martek's chewable DHA capsules containing 200mg in each capsule. The treatment will be provided as approximately 25mg/kg/day and 35mg/kg/day.
  These dosages will be divided BID-TID and will be given for 4 weeks.
  Other Names: Martek; DHA
  Arms: Docosahexanoic Acid Supplement
Dietary Supplement: Placebo — Placebo identical to active treatment.
  Arms: Placebo

SUMMARY:
Oral supplementation of patients affected by cystic fibrosis with docosahexanoic acid (DHA) will result in normalization of the known fatty acid derangements in these patients and will diminish the production of proinflammatory isoprostanes such as 8-isoprostane-PGF2α.

DETAILED DESCRIPTION:
The study design will be a single-center, randomized, placebo-controlled, cross-over trial. After informed consent has been obtained, 18 eligible subjects with pancreatic insufficient cystic fibrosis will be enrolled in the study. Participants will take part in two 4 week study sessions, each separated by a 4 week washout period. One session will involve treatment with placebo and the other two sessions will provide treatment with approximately 25mg and 35 mg of DHA/kg of body weight. The patients will be assigned to each of the treatment sessions in random order, as described above. The DHA source will be provided by Martek Biosciences Corporation, Columbia, MD, USA in the form of a chewable capsule containing 200 mg of DHA. The placebos will be identical to the DHA supplement but will not contain the active ingredient, DHA. Subjects will be instructed to take the study capsules in addition to their normal doses of pancreatic enzymes with meals and to maintain their usual diets. Blood, urine, and exhaled breath condensate samples will be collected at baseline and after completion of each of the study periods. Patients will be screened and enrolled when they present to clinic for their routine check-up. The subjects have routine blood work at their annual check-ups, and when possible will have an additional tube of blood saved for the baseline fatty acid profiles so as to avoid unnecessary blood draws. Following each study period, blood draw, urine collection, and exhaled breath condensate (EBC) will be collected at the Vanderbilt Clinical Research Center. The patients will also be given the supply of DHA and placebo (for the entire study) at time of enrollment. The order in which they take the supplement or the placebo will be determined using a randomization table.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on sweat chloride value > 60 mEq/L or genotyping
* Pancreatic insufficiency, defined by requirement for treatment with exogenous pancreatic enzymes
* FEV 1 > 40
* Less than 3 pulmonary exacerbations in the last year (as diagnosed by pulmonary attending physician)
* Age greater than 6 years
* Capability of performing pulmonary function tests
* Ability to swallow gel capsule
* Ability to comply with medication use, study visits, and study procedures
* Written informed consent obtained from subject or study subject's legal representative

Exclusion Criteria:

* Presence of severe CF-related liver disease, including SGOT or SGPT>3 times the normal limits, history of biliary cirrhosis, or portal hypertension
* Severe pulmonary disease, as defined by FEV1 < 40%
* Elevated serum creatinine or BUN
* Pregnancy
* PT >1.5 time normal
* Diabetes mellitus
* Daily use of NSAIDs or other anticoagulants
* History of fish allergy
* Use of ticlopidine, clopidogrel, dipyridamole
* Use of glucocorticoids
* History of lung transplant or currently on lung transplantation list
* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Exhaled breath 8-isoprostane-PGFα and urine 8-isoprostane-PGFα | 4 measurements: baseline and then one measurement after each of the three 4-week study periods

SECONDARY OUTCOMES:
Fatty acid profile analysis including esterification sites in plasma | 4 measurements - Baseline and then one measurement after each of the three 4-week study periods

CONTACTS AND LOCATIONS:
Overall Officials: Michael G O'Connor, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States